CLINICAL TRIAL: NCT04807192
Title: CMP-001 in Combination with Pre-Operative Stereotactic Body Radiation Therapy in Patients with Early Stage Triple Negative Breast Cancer: an Open-Label, Window of Opportunity, Randomized Phase 2 Clinical Study
Brief Title: CMP-001 and Pre-operative Stereotactic Body Radiation Therapy (SBRT) in Early Stage Triple Negative Breast Cancer (TNBC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr K. Zaman, MD, Medical director of the Breast Center at CHUV, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0009-CyberImmunoBreast
Record Dates: First submitted 2021-02-12; First posted 2021-03-19 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: SBRT (Experimental)
  Interventions: Radiation: stereotactic body radiotherapy
- Arm 2: CMP-001 + SBRT (Experimental)
  Interventions: Radiation: stereotactic body radiotherapy; Drug: CMP-001

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — one administration of SBRT 8 Gy at D1
Drug: CMP-001 — 4 sequential administrations of CMP001 at Day 1 (SC), Day 5 (±1) (IT), Day 9 (±1) (IT) and Day 16 (±1) (IT)
  Arms: Arm 2: CMP-001 + SBRT

SUMMARY:
This is an open-label, randomized, window-of-opportunity phase 2 clinical study evaluating the biological activity of preoperative Stereotactic Body RadioTherapy (SBRT) alone (Arm 1), and combined with subcutaneous (SC) followed by intra-tumoral (IT) administrations of CMP-001 (Arm 2), in subjects with early stage TNBC. Safety and efficacy of the treatments are also examined.

The main hypothesis that the study treatment induces an increase in stromal tumor infiltrating lymphocytes (sTILs) will be explored in each arm separately.

The study is designed as a randomized selection study, with randomization used to address patient selection bias while each arm is run as an independent study. No formal statistical comparison between the two arms is planned.

40 patients will be equally (1:1) randomized in this study (20 per arm), stratified into two groups according to primary treatment strategy (upfront surgery versus neoadjuvant chemotherapy).

DETAILED DESCRIPTION:
This is a Phase 2, proof of principle study that explores the therapeutic window between diagnosis and upfront surgery or start of the neoadjuvant chemotherapy in patients with early stage invasive TNBC.

The presence of tumor infiltrating lymphocytes (TILs) within the tumors of patients with early invasive TNBC has been associated with improved prognosis. The hypothesis of this study is that pre-operative stereotactic radiotherapy (SBRT) and SBRT combined with CpG (CMP-001), a Toll-like receptor (TLR) 9 agonist will induce an increase in stromal TILs (sTILs) in the tumor in patients with early invasive TNBC, which theoretically should improve those patients' prognosis.

There is growing evidence indicating that RT induces massive release of tumor-associated antigens (TAAs) during cancer cell death. RT enhances tumor immunogenicity and increases the presence of effector immune cells to the tumor site. It increases availability of tumor antigens and promotes antigen capture, cell migration to the lymph nodes, polarization towards a tolerogenic or immunogenic phenotype or migration of lymphocytes into the tumor. Doses of around 8 Gray (Gy) induce more important immune infiltration.

SBRT is a precise technique of irradiation within the tumor permitting high dose delivery in a safe manner with tight margins. In our study, the irradiated tissue will then be removed by surgery, allowing for standard of care irradiation to be administered postoperatively. However, the preoperative SBRT on the tumor might increase intratumoral or stromal TILs' presence.

CMP-001 (vidutolimod, CYT003, QbG10) has already been shown to increase CD8+ T cell intratumoral infiltration in early clinical data, and ongoing data of a phase Ib clinical trial combining intratumoral (IT) injections of CMP-001 (3-10 mg) in melanoma lesions with Pembrolizumab show rapid abscopal responses in other skin lesions after 3 injections. The combination of IT CMP-001 and SBRT, through increased TAA release and immunologic enhancement due to the TLR9 agonist, might ultimately result in a clinically meaningful " in-situ vaccination " effect through enhancement of the host's antitumor immunity, promoting immune eradication of micrometastatic disease. The TNBC population is prone to micrometastatic disease, even at early stages; therefore any of these experimental treatments might result in increased TILs' infiltration, which theoretically would bring potential benefits in distant control of the disease and overall survival improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Signed study Informed Consent Form prior to the initiation of any study procedures
2. Women age ≥18 years
3. Histologically confirmed diagnosis of triple negative breast cancer (TNBC) of early stage (cT1b-2, cN0-3b cM0) determined according to immunohistochemistry (IHC) / in situ hybridization (ISH). TNBC subtype is defined as:

   * Estrogen receptor (ER) <10%
   * Progesterone receptor (PR) <10%
   * Human epidermal growth factor receptor 2 (HER2) negative (not eligible for anti-HER2 therapy) defined as:

     * IHC 0, 1+ without ISH or
     * IHC 2+ and ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 6 signals/cells or
     * ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 6 signals/cells (without IHC)
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
5. Women with bilateral breast TNBC can be acceptable if both sides are TNBC (treatment is allowed to be administered to one breast only).
6. Capable of understanding and complying with protocol requirements
7. A planned breast surgery (Breast conserving surgery [BCS] or mastectomy) or neoadjuvant chemotherapy.
8. Presence of measurable disease in the breast, defined as a lesion that can be accurately measured in at least one dimension with conventional techniques (Magnetic resonance imaging [MRI] and/or ultrasound)
9. Primary tumor accessible to injections and biopsy. Multifocal and multicentric disease is allowed and the most accessible lesion will be injected. The lesion to be injected should be confined in a single irradiation volume that does not result in more than 30% of the whole breast.
10. The injected tumor should be located at least 5 mm from the skin or pectoral muscle
11. Most recent laboratory values (within 28 days prior to randomization) meet the following standards:

    1. Bone marrow function:

       * neutrophil count ≥1.5 G/L
       * hemoglobin ≥ 90 g/L
       * platelet count ≥ 100 G/L
    2. Liver function:

       * total bilirubin within normal ranges of each institution (except patients with Gilbert's syndrome who must have total bilirubin < 3.0 mg/dL)
       * aspartate aminotransferase (AST) ≤ 2.5 times the ULN range.
       * alanine aminotransferase (ALT) ≤ 2.5 times the ULN range
    3. Renal function: estimated glomerular filtration rate (eGFR) ≥ 40 ml/min/1.73 m2 (according to Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
12. For women of childbearing potential (WOCBP):

    1. Agreement to use an acceptable method of effective contraception from screening until 30 days after last study treatment (RT and CMP-001).
    2. WOCBP must have a negative urine/blood pregnancy test within 7 days before randomization. A positive urine test must be confirmed by a serum pregnancy test.

Exclusion Criteria:

Subjects presenting with any of the following do not qualify for entry into the study:

1. Breast-feeding women

   Medical history and concurrent diseases:
2. History of malignancy other than TNBC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma of the cervix in situ, non-melanoma skin carcinoma, ductal carcinoma in situ, or Stage I uterine cancer
3. Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
4. Developed autoimmune disorders of Grade 4 while on prior immunotherapy. Subjects who developed autoimmune disorders of Grade ≤ 3 may enroll if the disorder has resolved to Grade ≤ 1 and the subject has been off systemic steroids for at least 2 weeks.
5. Any concurrent uncontrolled illness, including mental illness or substance abuse, which in the opinion of the Investigator, would make the subject unable to cooperate and participate in the trial
6. Severe uncontrolled cardiac disease within 6 months before Screening, including but not limited to uncontrolled hypertension; unstable angina; myocardial infarction (MI) or cerebrovascular accident (CVA)
7. Active autoimmune disease:

   * Participants with well controlled asthma and/or mild allergic rhinitis (seasonal allergies) are eligible
   * Participants with the following disease conditions are also eligible:

     * Vitiligo
     * Type 1 diabetes mellitus
     * Residual hypothyroidism due to autoimmune condition only requiring hormone replacement
     * Psoriasis not requiring systemic treatment conditions not expected to recur in the absence of an external trigger are permitted to enroll
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to CMP-001
9. Any history of adrenal deficiency

   Prohibited treatments and/or therapies:
10. Any prior ipsilateral breast irradiation.
11. Received investigational therapy with another drug or biologic within 28 days prior to treatment study.
12. Require systemic pharmacologic doses of corticosteroids at or above the equivalent of 10 mg/day prednisone; replacement doses, topical, ophthalmologic and inhalational steroids are permitted. Subjects who are currently receiving steroids at a dose of < 10 mg/d do not need to discontinue steroids prior to randomization.
13. Requires prohibited treatment (i.e., non-protocol specified anticancer pharmacotherapy, surgery or conventional radiotherapy for treatment of malignant tumor).
14. For arm 2: Requires concomitant treatment with warfarin. Other anticoagulants (ie, low molecular weight heparins, non-steroidal anti-inflammatory drugs) are allowed as long as the institutional guidelines requiring their withholding for interventional radiology procedures can be followed.
15. Administration of a live, attenuated vaccine within 2 weeks before randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To assess and describe independently in each arm the biological activity (increase in sTILs) of CMP-001 combined with SBRT and of SBRT alone in patients with early stage TNBC in a preoperative setting | Evaluated between baseline and surgery (up to 7 weeks)
  A 10% increase in the presence of TILs (between baseline and surgery/biopsy before start of the neoadjuvant chemotherapy) is the defined threshold for efficacy.
  Percentage of sTILs will be quantified using hematoxylin and eosin (H&E) staining and immunohistochemistry (IHC) as per current consensus.

SECONDARY OUTCOMES:
Toxicity of CMP-001 combined with SBRT and of SBRT alone | (S)AEs collected continuously from the time of informed consent signature until end of treatment visit, which correspond to Day 51 to 60.
  Assessement of the incidence and severity of AEs and SAEs
Tumor response: pCR and pPR | evaluation at surgery (between day 21 and day 30 post-SBRT) or change from baseline to surgery (up to 7 weeks)
  Percentage of patients with a pathological complete response (pCR) and pathological Partial Response (pPR) for the patients with upfront surgery in the breast tumoral lesion(s) (lymph node tumoral lesion(s) not included)
Tumor response: residual tumor cells | evaluation at breast biopsy (between day 16 and day 30 post-SBRT)
  Estimated percentage of residual tumor cells in the breast and lymph node biopsies before the start of the neoadjuvant chemotherapy (for patients in the neoadjuvant group)
Tumor response: minimal residual cancer | evaluation at surgery (between day 21 and day 30 post-SBRT) or change from baseline to surgery (up to 7 weeks)
  Percentage of patients with minimal residual cancer as assessed by the residual cancer burden index (RCB) at upfront surgery in the breast tumoral lesion(s) (lymph node tumoral lesion(s) not included). The index will also be estimated in the biopsy done before the neoadjuvant chemotherapy of patients without upfront surgery.
Tumor response: Ki-67 | evaluation at surgery (between day 21 and day 30 post-SBRT) or change from baseline to surgery (up to 7 weeks)
  Mean change of proliferation index Ki-67 from baseline at upfront surgery / biopsy before the start of the neoadjuvant chemotherapy.
Tumor response: change in tumor characteristics | evaluation at surgery (between day 21 and day 30 post-SBRT) or change from baseline to surgery (up to 7 weeks)
  Mean change in tumor characteristics and peritumoral tissues as assessed by breast MRI and/or ultrasound (US) from baseline at upfront surgery / imaging before the start of the neoadjuvant chemotherapy. Data will also be compared to previously reported findings.
Time-to-event (TTE) | time from the date of randomization to the date of earliest objective tumor recurrence (up to 2 years from randomization)
  defined as time from the date of randomization to the date of earliest objective tumor recurrence, including progression that precludes surgery, or local or distant disease recurrence (deaths are censored)
Event-free survival (EFS) rate | at 24 months
  EFS rate is defined as the percentage of patients who are alive and without event (protocol-defined progression prior to surgery / start of the neoadjuvant chemotherapy; local, regional, or distant recurrence of breast cancer following curative surgery; a new breast cancer; another new onset malignancy; or death as a result of any cause) at month 24, per the Kaplan-Meier estimate of recurrence-free survival at 24 months.
Distant disease-free survival (DDFS) rate | at 24 months
  DDFS rate is defined as the percentage of patients without objective distant tumor recurrence (outside of the ipsilateral locoregional region) at month 24, per the Kaplan-Meier estimate of distant tumor recurrence-free survival at 24 months.
Overall survival (OS) rate | at 24 months
  OS rate is defined as the percentage of patients who are alive at month 24, per the Kaplan-Meier estimate of overall survival at 24 months (as event is considered the death from any cause).
Biological activity (difference between the 2 arms) | Evaluated between baseline and surgery for both arms (up to 7 weeks)
  sTILs increase will be compared between the two arms

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV Oncology Department, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No